CLINICAL TRIAL: NCT04512352
Title: A Large Scale Cross-sectional Survey and a Randomized Control Study on the Effectiveness of an Early Childhood Family-Based and Internet-Based Intervention
Brief Title: An Early Childhood Internet-based and Family-based Intervention Study
Acronym: ECII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: early-childhood-2020
Record Dates: First submitted 2020-05-15; First posted 2020-08-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2020-08

CONDITIONS: Early Childhood Development
Keywords: Social mobility & poverty; Internet & family-based; Early childhood intervetion; Intergenerational; Productive aging

STUDY DESIGN:
Intervention Model Description: Large-scale survey: Using the stratified sampling method, a randomized list of 60 samples was selected from the official list of 506 kindergartens-cum-child care center provided by the Bureau of Education. Out of the 60 schools, a total of 40 schools from 12 NGOs agreed to join the survey. As of April 2019, we have received 700 responses for the survey.
  Intervention Study: There are two phases of intervention in this stage. The total sample size for both phases is 200 parent-child dyads. For both phases, the team applied stratified randomization method for randomization. Participants were assigned to either treatment group or wait-list control group on a school basis.
Who Masked: Participant
Masking Description: Participants are not aware of which arm they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Online curriculum has been delivered to this group of participants on an Internet-based platform
  Interventions: Other: Online curriculum
- Wait-list control group (No Intervention): Participants in wait-list control group would not have access to the online curriculum until the intervention process for treatment group is finished.

INTERVENTIONS:
Other: Online curriculum — The psychologist and our advisory team had successfully developed a total of 100 hours of parenting curriculum.
  The adopted curriculum had focused on using play to facilitate parents in promoting their children's development in cognitive, motor, emotional and social aspects. Play-based activities are instrumental in improving children's development. Given that parents in poverty had difficulties spending time and money travelling back-and-forth to the training site and their homes, the research team decided to use e-learning as the medium of learning for our parenting programme. Web-based learning has the advantage of cutting time and travelling costs, which are luxuries to many parents in poverty.
  Arms: Treatment group

SUMMARY:
The poverty rate among children under 18 years old in Hong Kong in 2015 was 18% after social welfare intervention. James Heckman, a Nobel Prize winner in Economics, advocates early childhood investment to enhance social mobility, given its lifelong impact of on child development. However, few randomized control trails have been used to examine the effectiveness of early childhood intervention in promoting social mobility through child development in Hong Kong. To fill these gaps, we propose an interdisciplinary intervention study involving academics from economics, sociology, social work, gerontology, education, and psychology to investigate methods to promote the social mobility of children living in poverty through early intervention.

The overall objective is to enhance the developmental outcomes of children in poverty by utilizing parental resources within a family system, technological resources available in modern metropolis and the human resources enjoyed by the elderly in Hong Kong.

The primary objective is to evaluate an internet- and family-based intervention to promote the development of children in poverty enrolled in the first year of Hong Kong's nurseries, who are mostly aged 24 months to three years. The examined outcomes will be the developmental well-being of participating children and parenting attitudes and behaviors, with the long-term goal of promoting their social mobility to break the cycle of poverty. In the long run, we aim to establish the proposed intervention in policy to promote the development of disadvantaged children.

The secondary objective is to identify intergenerational volunteerism as a means for productive aging through a mentoring program using older adults as mentors to participating parents.

DETAILED DESCRIPTION:
The proposed research consists of three phases. The first phase will be a cross-sectional survey with a sample of 1,000 cases from 60 nurseries cum kindergartens to explore the family demographics and developmental profiles of low-income children in comparison to others. The second phase will be a randomized control trail implementing two waves of a 10-month internet-based intervention with 200 toddler-parents dyads from 20 to 30 of the original 60 nurseries. Interventions will be delivered by older mentors professionally trained by the research team. All children, parents and elderly mentors will be evaluated through a set of outcome measurements to assess the effectiveness of the program. The last phase will involve the dissemination of research information that may become building blocks for policies on internet-based early childhood education, poverty alleviation and social mobility enhancement, as well as productive aging.

ELIGIBILITY:
Inclusion Criteria:

* Parents who have children enrolled in the first year of Hong Kong nurseries ("N1"), mostly aged 24 months to 3 years

Exclusion Criteria:

* Parents who do not have children enrolled in the first year of Hong Kong nurseries ("N1")

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development- Third Edition | Change from baseline assessment at 10 months
  Bayley-III is a comprehensive tool to identify development issues during early childhood through direct assessment of the child. Domains include: Cognitive, Receptive Communication, Expressive Communication, Fine Motor, Gross Motor. The minimum scaled score is 1 and maximum scaled score is 19. A higher score means a better outcome.

SECONDARY OUTCOMES:
Parenting Sense of Competence Scale- Chinese | Change from baseline assessment at 10 months
  Parenting Sense of Competence Scale- Chinese (C-PSOC) was used to measure parenting sense of competence and satisfaction. The minimum score is 17 and the maximum score is 102. A higher score means a better outcome.
Chinese version of the Parental Feeding Style Questionnaire | Change from baseline assessment at 10 months
  A Chinese version of the parental feeding style questionnaire (PFSQ; Tam et al., 2014) was used, which covers: (1) instrumental feeding; (2) emotional feeding; (3) promoting and encouraging of feeding; and (4) control over children's eating. The minimum score is 27 and the maximum score is 135. A higher score means a better outcome.
Connor-Davidson Resilience Scale 10-item | Change from baseline assessment at 10 months
  Connor-Davidson Resilience Scale 10-item version (CD-RISC-10) was used to assess parents' resilience. The minimum score is 10 and the maximum score is 50. A higher score means a better outcome.
The Multidimensional Scale of Perceived Social Support-Chinese | Change from baseline assessment at 10 months
  The Multidimensional Scale of Perceived Social Support-Chinese Version (MSPSS-C) was used which measured the social support network of and support from friends, and perceived social support from family from parents' perspectives. The minimum score is 12 and the maximum score is 84. A higher score means a better outcome.

OTHER OUTCOMES:
The Ages and Stages Questionnaires (ASQ) -3 (Third Edition) | Change from baseline assessment at 10 months
  This scale is parent-reported and measures child development. It covers the following aspects: Communication, gross motor skills, fine motor skills, problem-solving, and personal-social skills. The minimum score is 0 and the maximum score is 300. A higher score means a better outcome.
Ages and Stages Questionnaire: Social-Emotional- 2 (Second Edition) | Change from baseline assessment at 10 months
  This scale is parent-reported and measures child development. This scale assesses social-emotional competence and challenging behaviors. The minimum score is 0 and the maximum score is 540. A higher score means a worse outcome.
Strengths and Difficulties Questionnaire | Change from baseline assessment at 10 months
  This scale is parent-reported and measures child development. It assesses parent's perception of children's behavioral problems, including emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships problem, and prosocial behavior. Each domain's minimum score is 0 and maximum is 10. For all domains except for prosocial behavior, a higher score means a worse outcome. For the prosocial behavior domain, a higher score means a better outcome.
Bayley Scales of Infant and Toddler Development- Third Edition: Social-Emotional | Change from baseline assessment at 10 months
  This scale is parent-reported and measures child development. Social-Emotional has 35 items. The minimum score is 0 and maximum score is 140. A higher score means a better outcome.
Bayley Scales of Infant and Toddler Development- Third Edition: Adaptive Behavior | Change from baseline assessment at 10 months
  This scale is parent-reported and measures child development. Adaptive Behavior includes 10 domains: Communication (25 items), Community Use (22-items), Functional Pre-Academics (23-items), Home Living (25-items), Health and Safety (24-items), Leisure (22-items), Self-Care (24-items), Self-Direction (25-items), Social (24-items), Motor Skills (27-items). The minimum score for the Adaptive Behavior composite is 0 and the maximum is 723. A higher score means a better outcome.
The General Functioning Subscale of the McMaster Family Assessment Device | Change from baseline assessment at 10 months
  The General Functioning Subscale of the McMaster Family Assessment Device (Epstein, Baldwin, and Bishop, 1983) was used to measure the family functioning. The minimum score is 12 and the maximum score is 48. The higher the score, the worse the outcome.
Parenting Stress Index - Short Form | Change from baseline assessment at 10 months
  PSI-SF was used to measure stress, which includes sub-scales: parental distress, parent-child dysfunctional interaction, and difficult child. The minimum score is 36 and the maximum score is 180. A higher score means a worse outcome.
The Depression, Anxiety and Stress Scale - 21 Items | Change from baseline assessment at 10 months
  DASS-21 was used to measure depression, anxiety and stress. The minimum score is 0 and the maximum score is 63. A higher score means a worse outcome.
Interpersonal Mindfulness in Parenting (IEMP) scale, Chinese version | Change from baseline assessment at 10 months
  IEMP was used to measure parental mindfulness, which has subscales: awareness & present-centered attention, non-judgment, and non-reactivity. The minimum score is 31 and the maximum score is 155. A higher score means a better outcome.
Psychological and Behavioral Control | Change from baseline assessment at 10 months
  This Chinese scale was originally developed by Dr. Daniel Shek (2006) and was adapted by the research team from adolescent-reported to parent-reported to assess levels of parental psychological control and behavioral control of their children. The minimum score is 23 and the maximum score is 92. The higher the score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Sung-Chan, Ph.D, Principal Investigator — Hong Kong Institute of Economics and Business Strategy
Locations (6):
- Hong Kong (6):
  - Hong Kong Christian Service, Hong Kong
  - Hong Kong Lutheran Social Service, Hong Kong
  - Hong Kong Young Women's Christian Association, Hong Kong
  - Po Leung Kuk, Hong Kong
  - The Salvation Army, Hong Kong
  - Tung Wah Group of Hospitals, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IPD shall be released ten years upon the completion of this project. For research purpose only, interested parties shall write to us to get the data.
Supporting Information: Analytic Code
Time Frame: Ten years upon the completion of this project
Access Criteria: For research purpose only